CLINICAL TRIAL: NCT02136992
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial for Clinical Efficacy and Safety of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Clinical Efficacy and Safety of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis
Acronym: IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Huiping Li, Huiping Li, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH01312
Record Dates: First submitted 2014-05-11; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (without active ingredient) (Placebo Comparator): placebo will be taken two tablets 3 times a day during the whole study process.
  Interventions: Drug: Pirfenidone; Drug: placebo
- Pirfenidone（200mg） (Experimental): Pirfenidone（200mg）tablets will be taken two tablets 3 times a day during the whole study process.
  Interventions: Drug: Pirfenidone; Drug: placebo

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone（200mg）tablets will be taken two tablets 3 times a day during the whole study process.
Drug: placebo — placebo will be taken two tablets 3 times a day during the whole study process

SUMMARY:
Pirfenidone as anti-fibrosis drug developed in recent years demonstrated the potential anti- fibrotic effect, but so far there were no domestic studies about pirfenidone's efficacy and safety evaluation in china. The aim of this study was to evaluate the efficacy and safety of pirfenidone in patients with idiopathic pulmonary fibrosis (IPF) through the observation of a large sample of clinical cases.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy and safety of pirfenidone in patients with idiopathic pulmonary fibrosis (IPF) through the observation of a large sample of clinical cases. During the observation, study visits will occur at the end of 12w, 24w, 36w, 48w.all participants will be required to check the various efficacy and safety indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed;
2. Age ≤75 years;
3. Clinically or multidisciplinary diagnosed idiopathic pulmonary fibrosis(see 2011 guidance );
4. Resting state PaO2≥50mg, FVC%≥45% normal predicted value and DLCO≥30% normal predicted value.

Exclusion Criteria:

1. Allergic to pirfenidone;
2. Patients with serious Significant pulmonary infection need anti-infection treatment;
3. Patients who has taken interferon, penicillamine or other agents for the treatment of IPF;
4. Patients who has taken prednisone(≥50mg) or other glucocorticoid in the past 1 month;
5. Patients who has taken immunosuppressants in the past 1 month;
6. Patients who has taken amiodarone which may cause pulmonary fibrosis in the past 3 months;
7. Patients with malignant tumor in the past 5 years;
8. Participated in other clinical trials in the past 3 months;
9. Patients with serious heart disease(NYHA class Ⅲ-Ⅳ), liver disease(ALT or AST 2 times above the upper level of normal value range), kidney disease(Cr above the upper level of normal value range);
10. Pregnant or lactating women;
11. The investigator assessed as inappropriate to participate in this clinical trial.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in forced vital capacity (FVC) | 48 weeks
  to evaluate changes in FVC from baseline to 12 weeks /24 weeks/36 weeks/48 weeks

SECONDARY OUTCOMES:
changes in lung function (including Forced expiratory volume in one second (FEV1) and The differences of diffusing capacity of the lung for carbon monoxide (DLco) ) | 48week
  Lung function will be measured as improved/stabilized/exacerbated from baseline to 12 weeks/24 weeks/36 weeks/48 weeks
Changes in 6 minute walk distance (6MWD) | 48 weeks
  Changes in 6 minute walk distance (6MWD) and from baseline to 12/24/36/48weeks
Life quality: assessed by St. George respiratory questionnaire (SGRQ). | 48 weeks
  Life quality will be assessed as improved if SGRQ single or total score increased >4% when completing the trial; Life quality will be assessed as stabilized if SGRQ single or total score changes within the range of 4% when completing the trial; Life quality will be assessed as exacerbated if SGRQ single or total score decreased >4% when completing the trial.
Dyspnea score according by Modified Medical Research Center(MMRC) | 48 weeks
  to measure rating dyspnea according by Medi Medical Research Center(MMRC)

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, Principal Investigator — Shanghai Pulmonary Hospital , Tongji University